CLINICAL TRIAL: NCT01584609
Title: A Randomized, Concurrent Controlled Trial to Assess the Safety and Effectiveness of the Separator 3D as a Component of the Penumbra System in the Revascularization of Large Vessel Occlusion in Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLP 4853; CLP 4853 (Other: Penumbrainc)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: ischemic stroke; large vessel occlusion; mechanical thrombectomy; revascularization; Penumbra System; Separator 3D
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Penumbra System with Separator 3D (Experimental)
  Interventions: Device: Penumbra System with Separator 3D
- Penumbra System alone (Active Comparator)
  Interventions: Device: Penumbra System alone

INTERVENTIONS:
Device: Penumbra System with Separator 3D — The Separator 3D is an additional Separator with a new tip configuration for the Penumbra System.
  Arms: Penumbra System with Separator 3D
Device: Penumbra System alone — The Penumbra System® is a new generation of neuro-embolectomy devices specifically designed to remove thrombus through aspiration.The treatment paradigm of this System involves the introduction of the Reperfusion Catheter through a guide catheter into the intracranial vasculature, and guided over an appropriate guidewire to the site of primary occlusion. The Reperfusion Catheter is used in parallel with the Separator and an aspiration source (Aspiration Pump) to separate the thrombus and aspirate it from the occluded vessel.
  Arms: Penumbra System alone

SUMMARY:
This is a prospective, randomized, single blind, concurrent controlled, multi-center study. Patients presenting with symptoms of acute ischemic stroke who have evidence of a large vessel (2.5mm or greater in diameter) occlusion in the cerebral circulation will be assigned to either the Penumbra System with the Separator 3D or the Penumbra System without the Separator 3D. Each treated patient will be followed and assessed for 3 months after randomization. Up to 230 evaluable patients at up to 50 centers presenting with acute ischemic stroke in vessels accessible to the Penumbra Separator 3D System for revascularization within 8 hours of symptom onset. The hypothesis to be tested is that the safety and effectiveness of the Penumbra System with the Separator 3D for the revascularization of large vessel occlusion is not inferior to the Penumbra System alone.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 85 years of age
* Present with symptoms consistent with an acute ischemic stroke for revascularization within 8 hours from symptom onset
* Refractory to or not eligible for IV rtPA therapy., e.g., presenting between 0 and 3 hours from symptom onset AND contraindicated for IV rtPA, or presenting between 3 and 8 hours of symptom onset, or evidence of persistent occlusion from vascular imaging after IV rtPA
* Evidence of a large vessel (2.5mm or greater in diameter) occlusion in the cerebral circulation
* NIH Stroke Scale (NIHSS) score 8 or more points
* Signed informed consent

Exclusion Criteria:

* History of stroke in the past 3 months.
* Females who are pregnant
* Pre-existing neurological or psychiatric disease that could confound the study results such as a pre-stroke mRS score 1 or higher
* Known severe allergy to contrast media
* Uncontrolled hypertension (defined as systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg)
* CT evidence of the following conditions at randomization:

  * Significant mass effect with midline shift
  * Large infarct region >1/3 of the middle cerebral artery territory
  * Evidence of intracranial hemorrhage
* Angiographic evidence of an arterial stenosis proximal to the occlusion that could prevent thrombus removal
* Angiographic evidence of preexisting arterial injury
* Rapidly improving neurological status prior to enrollment
* Bilateral stroke
* Intracranial tumors
* Known history of cerebral aneurysm or arteriovenous malformation
* Known hemorrhagic diathesis, coagulation deficiency, or on anticoagulant therapy with an International Normalized Ratio (INR) of >1.7
* Baseline platelets <50,000
* Use of IV heparin in the past 48 hours with PTT >1.5 times the normalized ratio
* Baseline glucose <50mg/dL or >300mg/dL
* Life expectancy less than 90 days prior to stroke onset
* Participation in another clinical investigation that could confound the evaluation of the study device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-04; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Frei, MD, Principal Investigator — Swedish Medical Center, Denver, CO
Locations (8):
- United States (8):
  - Hoag Hospital, Newport Beach, California
  - Swedish Medical Center, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Grady Health System, Atlanta, Georgia
  - St. Joseph Hospital- Healtheast, Saint Paul, Minnesota
  - Kaleida Health, Buffalo, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Derived] Nogueira RG, Frei D, Kirmani JF, Zaidat O, Lopes D, Turk AS 3rd, Heck D, Mason B, Haussen DC, Levy EI, Mehta S, Lazzaro M, Chen M, Dorfler A, Yoo AJ, Derdeyn CP, Schwamm L, Langer D, Siddiqui A; Penumbra Separator 3D Investigators. Safety and Efficacy of a 3-Dimensional Stent Retriever With Aspiration-Based Thrombectomy vs Aspiration-Based Thrombectomy Alone in Acute Ischemic Stroke Intervention: A Randomized Clinical Trial. JAMA Neurol. 2018 Mar 1;75(3):304-311. doi: 10.1001/jamaneurol.2017.3967. PMID 29296999

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Started | 98 | 100
Completed | 86 | 96
Not Completed | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (13.6) | 66.5 (12.5) | 66.9 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 54 | 111
  Male | 41 | 46 | 87
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 100 | 198

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Angiographic Revascularization of the Occluded Target Vessel
Description: Number of Participants with Angiographic revascularization of the occluded target vessel defined by mTICI grade 2-3
Time Frame: At immediate post-procedure
Population: Analysis population demonstrate outcomes of number of subjects that met endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 94 | 96
Participants | 82 | 79

2. Primary Outcome: Number of Device-related Serious Adverse Events
Time Frame: Within 24 hours post-procedure
Measure: Number; unit: Device-Related Serious Adverse Events
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 98 | 100
Device-Related Serious Adverse Events | 4 | 5

3. Primary Outcome: Number of Procedure-related Serious Adverse Event
Time Frame: Within 24 hours post-procedure
Measure: Number; unit: Procedure-related Serious Adverse Events
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 98 | 100
Procedure-related Serious Adverse Events | 10 | 14

4. Secondary Outcome: Good Clinical Outcome at 30 Days
Description: Defined by a 10 points or more improvement in the NIHSS at Discharge, a NIHSS score of 0-1 at Discharge; or a 30-day mRS score of 0-2. The NIHSS is a stroke scale that measures impairment caused by stroke. The Modified Rankin scale (mRS) measures neurological disability or dependence for stroke patients.
Time Frame: 30 days post-procedure
Population: Analysis population demonstrate outcomes of number of subjects that met endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 97 | 100
Participants | 58 | 55

5. Secondary Outcome: Number of Participants With 90 Day mRS Score 0-2
Time Frame: at 90 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 86 | 96
Participants | 39 | 44

6. Secondary Outcome: All Cause Mortality
Time Frame: At 90 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 98 | 100
Participants | 19 | 26

7. Secondary Outcome: Number of Symptomatic Intracranial Hemorrhage
Time Frame: Within 24 hours post-procedure
Measure: Number; unit: Symptomatic Intracranial Hemorrhage
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 98 | 100
Symptomatic Intracranial Hemorrhage | 3 | 5

8. Secondary Outcome: Good Neurological Outcome at 90 Days
Description: Defined by an mRS score of 0-2, or equal to the pre-stroke mRS score if the pre-stroke mRS score was higher than 2, or an improvement of 10 or more points on the NIHSS score
Time Frame: At 90 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
Number analyzed (Participants) | 86 | 96
Participants | 56 | 55

ADVERSE EVENTS:
Time Frame: Procedure up to 90 days
Description: Serious Adverse Events and Other (Not Including Serious): the total number of subjects analyzed is per protocol population. Data includes roll-in subjects and adjudicated by CEC. Events labeled as is in our Instructions for Use.
Arm/Group | Penumbra System With Separator 3D | Penumbra System Alone
All-Cause Mortality (participants affected / at risk) | 19/98 | 26/100
Serious Adverse Events (participants affected / at risk) | 38/88 | 49/93
Other Adverse Events (participants affected / at risk) | 81/88 | 83/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Penumbra System With Separator 3D (N=88) | Penumbra System Alone (N=93)
Nervous system disorders (Nervous system disorders) | 19 (19) | 28 (28)
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (11)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (8) | 10
Cardiac disorders (Cardiac disorders) | 10 (10) | 7 (7)
Vascular disorders (Vascular disorders) | 1 (1) | 9 (9)
Infections and infestations (Infections and infestations) | 2 (2) | 6 (6)
Renal and urinary disorders (Renal and urinary disorders) | 4 (4) | 1 (1)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 | 2
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Endocrine disorders (Endocrine disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions (General disorders) | 1 | 0
Immune system disorders (Immune system disorders) | 0 (0) | 1 (1)
Investigations (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Penumbra System With Separator 3D (N=88) | Penumbra System Alone (N=93)
Nervous System Disorders (Nervous system disorders) | 48 (48) | 59 (59)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 27 (27) | 30 (30)
Infections and Infestations (Infections and infestations) | 28 (28) | 25 (25)
Vascular Disorder (Vascular disorders) | 27 (27) | 25 (25)
Cardiac Disorders (Cardiac disorders) | 28 (28) | 23 (23)
Gastrointestinal Disorders (Gastrointestinal disorders) | 21 (21) | 29 (29)
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 24 (24)
General disorders and administration site conditions (General disorders) | 25 (25) | 20 (20)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 24 (24) | 19 (19)
Psychiatric disorders (Psychiatric disorders) | 14 (14) | 19 (19)
Renal and urinary disorders (Renal and urinary disorders) | 14 (14) | 12 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 10 (10) | 9 (9)
Investigations (Investigations) | 13 (13) | 6 (6)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2012-06-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT01584609/Prot_000.pdf
  • Statistical Analysis Plan (2013-02-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT01584609/SAP_001.pdf